CLINICAL TRIAL: NCT01940107
Title: Domiciliary Physiotherapy in Women Undergoing Treatment for Breast Cancer Radiation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Helio Carrara, MD, PhD, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: hhacarra
Record Dates: First submitted 2013-09-06; First posted 2013-09-11 (Estimated); Last update posted 2013-09-11 (Estimated); Status verified 2013-09

CONDITIONS: Frozen Shoulder,; Shoulder Pain
Keywords: breast cancer,; radiotherapy,; physical therapy,; upper limb
MeSH Terms: conditions — Bursitis; Shoulder Pain; Breast Neoplasms

ARMS (2):
- Control Group (CG) (Other): Control Group, which were subjected only to evaluations and to no exercise
  Interventions: Other: evaluations
- Study Group (SG) (Experimental): Study group (SG), was oriented to perform domiciliary exercises for the upper limbs.
  Interventions: Procedure: Protocol of physiotherapy exercises

INTERVENTIONS:
Other: evaluations — Only evaluations
  Arms: Control Group (CG)
Procedure: Protocol of physiotherapy exercises — Oriented domiciliary physiotherapeutic exercises
  Arms: Study Group (SG)

SUMMARY:
To observe the effect of domiciliary physiotherapy on the upper limb applied during the period of radiotherapy in women submitted to surgical and radiotherapy for breast cancer. The parameters evaluated were: shoulder range of movement (ROM) and arm circumference. There was significant difference between the ipsilateral and contralateral limbs for flexion, abduction and external rotation. There was no difference in perimetry in either group

ELIGIBILITY:
Inclusion Criteria:

* be diagnosed with unilateral breast cancer;
* be submitted to surgical and radiation treatment as part of the treatment for breast cancer.

Exclusion Criteria:

* patients with neurological or orthopedic diseases that could impair the upper limb movements
* bilateral breast cancer;
* prior thoracic radiotherapy;
* presence of distant metastasis.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-08; Primary Completion 2012-07 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Recovery of shoulder range of movements (ROM) and prevention of arm lymphedema | 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas de Ribeirão Preto da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo, Ribeirão Preto, Saõ Paulo, Brazil